CLINICAL TRIAL: NCT05129592
Title: A Randomized Controlled Trial Testing the Efficacy of Brief Messages to Correct Misperceptions About Nicotine
Brief Title: Can Exposure to Brief Messages Correct Misperceptions?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Other
Other Study IDs: 00015120A
Record Dates: First submitted 2021-10-01; First posted 2021-11-22 (Actual); Results first posted 2024-03-12 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Beliefs

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to view one of four messages. The message conditions are as follows: condition 1 will not contain either component of coherence; condition 2 will contain one element of coherence (a causal explanation for why the corrective information is accurate); condition 3 will contain the other element of coherence (an explanation for why the misinformation came to be believed); condition 4 will include both elements of coherence.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Nicotine corrective control (Active Comparator): A factual message about nicotine that does not contain a causal explanation for what actually causes tobacco-caused disease or an explanation for why the misperception that nicotine causes cancer may have come to be believed.
  Interventions: Behavioral: Coherent corrective messages
- Nicotine corrective with causal explanation (Experimental): A factual message about nicotine that contain a causal explanation for what actually causes tobacco-caused disease: tar and chemicals created in tobacco smoke when tobacco is lit on fire.
  Interventions: Behavioral: Coherent corrective messages
- Nicotine corrective with reason for misperception (Experimental): A factual message about nicotine that contains an explanation for why the misperception may have come to be believed: that health messaging often discuses nicotine and tobacco-caused disease at the same time and people incorrectly make the connection that nicotine causes cancer.
  Interventions: Behavioral: Coherent corrective messages
- Nicotine corrective with both components of coherence (Experimental): A factual message about nicotine that contains both a causal explanation for what actually causes tobacco-caused disease and an explanation for why the misperception may have come to be believed.
  Interventions: Behavioral: Coherent corrective messages

INTERVENTIONS:
Behavioral: Coherent corrective messages — Participants will be randomized to one of four message conditions: condition 1 will not contain either component of the coherence; condition 2 will contain one element of coherence (a causal explanation for why the corrective information is accurate); condition 3 will contain the other element of coherence (an explanation for why the misinformation came to be believed); condition 4 will include both elements of coherence.

SUMMARY:
This study seeks to assess the efficacy of educational messages to correct misperceptions. A large proportion of the American population incorrectly believes that nicotine is the chemical responsible for causing cancer in tobacco products.1-3 This misconception may reduce the likelihood that established smokers who are unwilling or unable to quit tobacco product use completely will switch to less harmful non-combustible products. An online experiment will be used to test if corrective messages can reduce this misperception. The experiment will also test the effects of messages on beliefs about the relative harms of other tobacco products discussed in the message and accuracy of inferential beliefs. This will be accomplished by asking participants questions about two tobacco products that are not explicitly discussed in the messages. The experiment will test if the two components of "narrative coherence," a concept identified in previous reviews of misperception correction as effective,4-6 is effective at reducing misperceptions about nicotine. Component 1 provides an explanation for why the new information is correct and component 2 provides an explanation for how the false information came to be believed. This study will use a factorial design to test the efficacy of the component of coherence individually as well as together. Hypotheses and Research Questions:

RQ1: Will participants exposed to different corrective message conditions differ in increased accuracy of beliefs (a) that nicotine does not cause cancer, (b) regarding the relative risk of e-cigarettes compared to cigarettes, (c) regarding the relative risk of very low nicotine cigarettes (VLNC) compared to cigarettes and (d) regarding the relative risk of nicotine replacement therapy compared to cigarettes.

H1: Participants exposed to the nicotine corrective message with both components of coherence will be significantly more likely to increase accuracy of beliefs regarding the relative harms of (a) smokeless tobacco compared to cigarettes and (b) cigarillos relative to cigarettes compared to those exposed to messages with just one component or no components of coherence.

H2: Participants exposed to the nicotine corrective message with both components of coherence will be significantly more likely to increase their intention to switch completely to a noncombustible product compared to those exposed to messages with just one component or no components of coherence.

ELIGIBILITY:
Inclusion Criteria:

* Are established smokers (have smoked at least 100 cigarettes in their lifetime and currently smoke some or all days)
* Are 21 years of age or older (the legal age of tobacco purchase in the US)
* Have not completed the cognitive interview during message pre-testing.
* Rate their agreement with the following statement as at least 50 out of 100: "To what extent do you agree with the following statement: The substance nicotine causes cancer."
* Are registered with MTurk in the United States.
* Have completed >= 5,000 HIITs within the MTurk system
* Have a HIIT approval rating of >= 97%

Exclusion Criteria:

* Are not established smokers
* Are younger than 21 years of age
* Participated in cognitive interviews during message pre-testing
* Are not registered with MTurk in the US
* Have completed < 5,000 HIITS
* Have a HIIT approval rating of <97%
* Rate their agreement with the following statement as less than 50 out of 100: "To what extent do you agree with the following statement: The substance nicotine causes cancer."

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 193 (Actual)
Dates: Start 2021-11-22 (Actual); Primary Completion 2022-01-30 (Actual); Study Completion 2022-08-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Meghan B Moran, PhD, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (1):
- Johns Hopkins Bloomberg School of Public Health, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Upon request, deidentified participant data collected during the study may be shared. Upon request, the PI may also share the study protocol, survey, and informed consent form. Data will be made available upon request beginning 3 months following publication of the final article from this study, with no end date. Data will be made available for analyses deemed appropriate by the study PI. Proposals should be directed to mmoran22@jhu.edu. Data requestors will need to sign a data access agreement.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 3 months following publication of the final article from this study

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Online recruitment began November 22, 2021 using Amazon Mechanical Turk. Funds to compensate participants were exhausted on November 23, 2021. An administrative delay in transferring funding created a delay in further recruitment, which was restarted on January 25, 2022 and was completed January 27, 2022.
Period: Overall Study
Arm/Group | Nicotine Corrective Control | Nicotine Corrective With Causal Explanation | Nicotine Corrective With Reason for Misperception | Nicotine Corrective With Both Components of Coherence
Started | 42 | 53 | 56 | 42
Completed | 42 | 53 | 56 | 42
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Nicotine Corrective Control | Nicotine Corrective With Causal Explanation | Nicotine Corrective With Reason for Misperception | Nicotine Corrective With Both Components of Coherence | Total
Number analyzed (Participants) | 42 | 53 | 56 | 42 | 193
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 39.5 [33 to 48] | 39 [32 to 55] | 40 [34.5 to 50] | 40.5 [33 to 51] | 40 [33 to 50]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 22 | 30 | 16 | 95
  Male | 15 | 31 | 26 | 26 | 98
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Non-Hispanic White | 33 | 46 | 44 | 33 | 156
  Ethnic/racial minority | 9 | 7 | 12 | 9 | 37
E-cigarette use [Count of Participants; unit: Participants]
  Current use (past 30-day use) | 12 | 13 | 19 | 11 | 55
  Ever use (not past 30 days) | 24 | 32 | 29 | 24 | 109
  Never use | 6 | 8 | 8 | 7 | 29
Self-reported very low nicotine cigarette use [Count of Participants; unit: Participants]
  Current use (past 30 days) | 3 | 1 | 2 | 2 | 8
  Ever use (not past 30 days) | 5 | 7 | 9 | 7 | 28
  Never use | 34 | 45 | 45 | 33 | 157
Smokeless tobacco use [Count of Participants; unit: Participants]
  Current use (past 30 days) | 3 | 2 | 1 | 3 | 9
  Ever use (not past 30 days) | 13 | 25 | 20 | 17 | 75
  Never use | 26 | 26 | 35 | 22 | 109
Nicotine replacement therapy use [Count of Participants; unit: Participants]
  Current use (past 30 days) | 8 | 4 | 6 | 6 | 24
  Ever use (not past 30 days) | 16 | 20 | 23 | 15 | 74
  Never use | 18 | 29 | 27 | 21 | 95
Cigarillo use [Count of Participants; unit: Participants]
  Current use (past 30 days) | 5 | 10 | 7 | 9 | 31
  Ever use (not past 30 days) | 19 | 26 | 28 | 24 | 97
  Never use | 18 | 17 | 21 | 9 | 65

OUTCOME MEASURES:

1. Primary Outcome: Change in Accuracy of Belief That Nicotine Causes Cancer
Description: The extent to which participants agree or disagree with the following statement: The substance nicotine causes cancer. Response options are a continuous scale from 0 "I do not agree at all" to 100, "I completely agree."
Time Frame: Baseline and up to 5 minutes after receiving the corrective message
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Nicotine Corrective Control | Nicotine Corrective With Causal Explanation | Nicotine Corrective With Reason for Misperception | Nicotine Corrective With Both Components of Coherence
Number analyzed (Participants) | 42 | 53 | 56 | 42
units on a scale | 52.6 (31.9) | 54.0 (35.3) | 39.2 (34.1) | 36.1 (35.4)
Statistical Analysis 1: Comparison: Nicotine Corrective Control vs Nicotine Corrective With Both Components of Coherence; Test type: Superiority; p = 0.095, ANCOVA — Sidak's adjusted p-value contrasting marginal linear predictions for the Nicotine corrective control and Nicotine corrective with both components of coherence; Controlling for baseline nicotine misperception (df=4); Mean Difference (Final Values) = 15.71, 95% CI 2-sided [-1.87 to 33.30], Standard Error of Mean 7.30 — Comparing Nicotine corrective control to the Nicotine corrective with both components of coherence
Statistical Analysis 2: Comparison: Nicotine Corrective With Causal Explanation vs Nicotine Corrective With Both Components of Coherence; Sidak's adjusted p-value contrasting marginal linear predictions for the Nicotine corrective with causal explanation and Nicotine corrective with both components of coherence; Test type: Superiority; p = 0.022, ANCOVA — Sidak's adjustment for multiple comparisons; Controlling for baseline nicotine misperception (df=4); Mean Difference (Final Values) = 18.67, 95% CI 2-sided [2.02 to 35.33], Standard Error of Mean 7.30 — Comparing Nicotine corrective control to the Nicotine corrective with both components of coherence
Statistical Analysis 3: Comparison: Nicotine Corrective With Reason for Misperception vs Nicotine Corrective With Both Components of Coherence; Sidak's adjusted p-value contrasting marginal linear predictions for the Nicotine corrective with reason for misperception and Nicotine corrective with both components of coherence; Test type: Superiority; p = 0.931, ANCOVA — Sidak's adjustment for multiple comparisons; Controlling for baseline nicotine misperception (df=4); Mean Difference (Final Values) = 3.69, 95% CI 2-sided [-12.76 to 20.15], Standard Error of Mean 7.30 — Comparing Nicotine corrective with reason for misperception to the Nicotine corrective with both components of coherence

2. Primary Outcome: Change in Relative Harm Beliefs Regarding E-cigarettes
Description: "The next questions are about electronic cigarettes. You may also know them as e-cigarettes, vapes, vape pens, mods, or by brand names like Juul, Suorin, SMOK, Fin, NJOY, Blu, e-Go, or Vuse. Some look like cigarettes, and others look like small boxes, pens, or pipes. From now on, we will refer to these products as e-cigarettes. E-cigarettes heat up a liquid to aerosolize it so people can inhale it. Although some e-liquid does not contain nicotine, we are only interested in e-cigarettes that DO contain nicotine. Please answer the following questions about e-cigarettes that contain nicotine." Response options are, "Much less harmful," "Somewhat less harmful," "Not less or more harmful," "Somewhat more harmful," "Much more harmful." Response options were dichotomized to low relative harm perceptions (much less harmful, somewhat less harmful) and high relative harm perceptions (much more harmful, somewhat more harmful, not less or more harmful).
Time Frame: Baseline and up to 5 minutes after receiving the corrective message
Measure: Count of Participants; unit: Participants
Arm/Group | Nicotine Corrective Control | Nicotine Corrective With Causal Explanation | Nicotine Corrective With Reason for Misperception | Nicotine Corrective With Both Components of Coherence
Number analyzed (Participants) | 42 | 53 | 56 | 42
Participants
  Low relative harm perception | 34 | 43 | 38 | 31
  High relative harm perception | 6 | 9 | 16 | 10
  Missing | 2 | 1 | 2 | 1
Statistical Analysis 1: Comparison: Nicotine Corrective With Causal Explanation vs Nicotine Corrective With Both Components of Coherence; Unadjusted logistic regression showing the effect of condition (Nicotine corrective with causal explanation compared to the Nicotine corrective with both components of coherence (reference group)) on e-cigarette relative harm beliefs; Test type: Superiority; p = 0.402, Regression, Logistic; Odds Ratio (OR) = 1.54, 95% CI 2-sided [0.56 to 4.24] — Odds of believing e-cigarettes are less harmful than cigarettes in the Nicotine corrective with causal explanation/odds of believing e-cigarettes are less harmful than cigarettes in the condition with both component of coherence
Statistical Analysis 2: Comparison: Nicotine Corrective Control vs Nicotine Corrective With Both Components of Coherence; Unadjusted logistic regression showing the effect of condition (Nicotine corrective control compared to the Nicotine corrective with both components of coherence (reference group)) on e-cigarette relative harm beliefs; Test type: Superiority; p = 0.292, Regression, Logistic; Odds Ratio (OR) = 1.83, 95% CI 2-sided [0.59 to 5.62] — Odds of believing e-cigarettes are somewhat or much less harmful than cigarettes in the control condition/odds of believing e-cigarettes are somewhat or much less harmful than cigarettes in the condition with both component of coherence
Statistical Analysis 3: Comparison: Nicotine Corrective With Reason for Misperception vs Nicotine Corrective With Both Components of Coherence; Unadjusted logistic regression showing the effect of condition (Nicotine corrective with reason for misperception compared to the Nicotine corrective with both components of coherence (reference group)) on e-cigarette relative harm beliefs; Test type: Superiority; p = 0.571, Regression, Logistic; Odds Ratio (OR) = 0.77, 95% CI 2-sided [0.30 to 1.93] — Odds of believing e-cigarettes are less harmful than cigarettes in the Nicotine corrective with reason for misperception/odds of believing e-cigarettes are less harmful than cigarettes in the condition with both component of coherence
Statistical Analysis 4: Comparison: Nicotine Corrective Control vs Nicotine Corrective With Both Components of Coherence; Adjusted logistic regression showing the effect of condition (Nicotine corrective control compared to the Nicotine corrective with both components of coherence (reference group)) on e-cigarette relative harm beliefs controlling for baseline beliefs and e-cigarette use; Test type: Superiority; p = 0.349, Regression, Logistic; Odds Ratio (OR) = 1.98, 95% CI 2-sided [0.47 to 8.26], Standard Error of Mean 1.44 — Odds of believing e-cigarettes are less harmful than cigarettes in the control condition/odds of believing e-cigarettes are less harmful than cigarettes in the condition with both component of coherence
Statistical Analysis 5: Comparison: Nicotine Corrective With Causal Explanation vs Nicotine Corrective With Both Components of Coherence; Adjusted logistic regression showing the effect of condition (Nicotine corrective with causal explanation compared to the Nicotine corrective with both components of coherence (reference group)) on e-cigarette relative harm beliefs controlling for baseline beliefs and e-cigarette use; Test type: Superiority; p = 0.355, Regression, Logistic; Odds Ratio (OR) = 1.76, 95% CI 2-sided [0.53 to 5.81], Standard Error of Mean 1.07 — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 6: Comparison: Nicotine Corrective With Reason for Misperception vs Nicotine Corrective With Both Components of Coherence; Adjusted logistic regression showing the effect of condition (Nicotine corrective with reason for misperception compared to the Nicotine corrective with both components of coherence (reference group)) on e-cigarette relative harm beliefs controlling for baseline beliefs and e-cigarette use; Test type: Superiority; p = 0.591, Regression, Logistic; Odds Ratio (OR) = 0.74, 95% CI 2-sided [0.24 to 2.25], Standard Error of Mean .42 — [estimate comment as in outcome 2, analysis 3]

3. Primary Outcome: Change in Relative Harm Beliefs Regarding NRT
Description: Participants will be shown a written description of NRT before answering questions about them: "The next questions are about nicotine replacement therapy (NRT). NRT is a medicine that is available as skin patches, chewing gum, nasal and oral sprays, inhalers, lozenges and tablets and delivers nicotine to the body. Nicotine replacement therapy is approved to help people quit smoking." Participants will also see a picture of these products with the description. Response options are, "Much less harmful," "Somewhat less harmful," "Not less or more harmful," "Somewhat more harmful," "Much more harmful." Response options were dichotomized to low relative harm perceptions (much less harmful, somewhat less harmful) and high relative harm perceptions (much more harmful, somewhat more harmful, not less or more harmful).
Time Frame: Baseline and up to 5 minutes after receiving the corrective message
Measure: Count of Participants; unit: Participants
Arm/Group | Nicotine Corrective Control | Nicotine Corrective With Causal Explanation | Nicotine Corrective With Reason for Misperception | Nicotine Corrective With Both Components of Coherence
Number analyzed (Participants) | 41 | 52 | 53 | 42
Participants
  Low relative harm perception | 39 | 47 | 50 | 40
  High relative harm perception | 2 | 5 | 3 | 2
Statistical Analysis 1: Comparison: Nicotine Corrective Control vs Nicotine Corrective With Both Components of Coherence; Test type: Superiority — Unadjusted logistic regression showing the effect of condition (Nicotine corrective control compared to the Nicotine corrective with both components of coherence (reference group)) on NRT relative harm beliefs; p = 0.980, Regression, Logistic; Odds Ratio (OR) = 0.98, 95% CI 2-sided [0.13 to 7.27], Standard Error of Mean .99 — Odds of believing NRT is less harmful than cigarettes in the control condition/odds of believing NRT is less harmful than cigarettes in the condition with both component of coherence
Statistical Analysis 2: Comparison: Nicotine Corrective With Causal Explanation vs Nicotine Corrective With Both Components of Coherence; Unadjusted logistic regression showing the effect of condition (Nicotine corrective with causal explanation compared to the Nicotine corrective with both components of coherence (reference group)) on NRT relative harm beliefs; Test type: Superiority; p = 0.382, Regression, Logistic; Odds Ratio (OR) = 0.47, 95% CI 2-sided [0.09 to 2.56], Standard Error of Mean .41 — Odds of believing NRT is less harmful than cigarettes in the Nicotine corrective with causal explanation/odds of believing NRT is less harmful than cigarettes in the condition with both component of coherence
Statistical Analysis 3: Comparison: Nicotine Corrective With Reason for Misperception vs Nicotine Corrective With Both Components of Coherence; Unadjusted logistic regression showing the effect of condition (Nicotine corrective with reason for misperception compared to the Nicotine corrective with both components of coherence (reference group)) on NRT relative harm beliefs; Test type: Superiority; p = 0.846, Regression, Logistic; Odds Ratio, log = 0.83, 95% CI 2-sided [0.13 to 5.23], Standard Error of Mean .79 — Odds of believing NRT is less harmful than cigarettes in the Nicotine corrective with reason for misperception/odds of believing NRT is less harmful than cigarettes in the condition with both component of coherence
Statistical Analysis 4: Comparison: Nicotine Corrective Control vs Nicotine Corrective With Both Components of Coherence; Adjusted logistic regression showing the effect of condition (Nicotine corrective control compared to the Nicotine corrective with both components of coherence (reference group)) on NRT relative harm beliefs controlling for NRT use; Test type: Superiority; p = 0.990, Regression, Logistic; Odds Ratio (OR) = 1.01, 95% CI 2-sided [0.13 to 7.74], Standard Error of Mean 1.05 — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 5: Comparison: Nicotine Corrective With Causal Explanation vs Nicotine Corrective With Both Components of Coherence; Adjusted logistic regression showing the effect of condition (Nicotine corrective with causal explanation compared to the Nicotine corrective with both components of coherence (reference group)) on NRT relative harm beliefs controlling for NRT use; Test type: Superiority; p = 0.458, Regression, Logistic; Odds Ratio (OR) = 0.51, 95% CI 2-sided [0.09 to 3.01], Standard Error of Mean .46 — [estimate comment as in outcome 3, analysis 2]
Statistical Analysis 6: Comparison: Nicotine Corrective With Reason for Misperception vs Nicotine Corrective With Both Components of Coherence; Adjusted logistic regression showing the effect of condition (Nicotine corrective with reason for misperception compared to the Nicotine corrective with both components of coherence (reference group)) on NRT relative harm beliefs controlling for NRT use; Test type: Superiority; p = 0.754, Regression, Logistic; Odds Ratio (OR) = 0.74, 95% CI 2-sided [0.12 to 4.76], Standard Error of Mean .70 — [estimate comment as in outcome 3, analysis 3]

4. Primary Outcome: Change in Relative Harm Beliefs Regarding Very Low Nicotine Cigarettes
Description: Participants will be shown a written description of very low nicotine cigarettes before answering questions about them: "The next questions are about very low nicotine cigarettes. A very low nicotine cigarette is a tobacco cigarette that is still smoked but has the vast majority (95% or more) of the nicotine removed from it. The average regular cigarettes typically contains 12-13 mg of nicotine. A very low nicotine cigarette could have less than 1 mg of nicotine in it. Very low nicotine cigarettes do not contain enough nicotine to maintain a physiological addiction to nicotine. Quest and Moonlight are brands of very low nicotine cigarettes." Participants will also see a picture of these products with the description. Response options were dichotomized to low relative harm perceptions (much less harmful, somewhat less harmful) and high relative harm perceptions (much more harmful, somewhat more harmful, not less or more harmful).
Time Frame: Baseline and up to 5 minutes after receiving the corrective message
Measure: Count of Participants; unit: Participants
Arm/Group | Nicotine Corrective Control | Nicotine Corrective With Causal Explanation | Nicotine Corrective With Reason for Misperception | Nicotine Corrective With Both Components of Coherence
Number analyzed (Participants) | 42 | 53 | 56 | 42
Participants
  Low relative harm perception | 28 | 30 | 25 | 23
  High relative harm perception | 13 | 23 | 29 | 18
  Missing | 1 | 0 | 2 | 1
Statistical Analysis 1: Comparison: Nicotine Corrective Control vs Nicotine Corrective With Both Components of Coherence; Unadjusted logistic regression showing the effect of condition (Nicotine corrective control compared to the Nicotine corrective with both components of coherence (reference group)) on VLNC relative harm beliefs; Test type: Superiority; p = 0.256, Regression, Logistic; Odds Ratio, log = 1.69, 95% CI 2-sided [0.68 to 4.15], Standard Error of Mean .78 — Odds of believing VLNC are less harmful than cigarettes in the control condition/odds of believing VLNC are less harmful than cigarettes in the condition with both component of coherence
Statistical Analysis 2: Comparison: Nicotine Corrective With Causal Explanation vs Nicotine Corrective With Both Components of Coherence; Unadjusted logistic regression showing the effect of condition (Nicotine corrective with causal explanation compared to the Nicotine corrective with both components of coherence (reference group)) on VLNC relative harm beliefs; Test type: Superiority; p = 0.961, Regression, Logistic; Odds Ratio (OR) = 1.02, 95% CI 2-sided [0.45 to 2.32], Standard Error of Mean .43 — Odds of believing VLNC are less harmful than cigarettes in the Nicotine corrective with causal explanation/odds of believing VLNC are less harmful than cigarettes in the condition with both component of coherence
Statistical Analysis 3: Comparison: Nicotine Corrective With Reason for Misperception vs Nicotine Corrective With Both Components of Coherence; Unadjusted logistic regression showing the effect of condition (Nicotine corrective with reason for misperception compared to the Nicotine corrective with both components of coherence (reference group)) on VLNC relative harm beliefs; Test type: Superiority; p = 0.345, Regression, Logistic; Odds Ratio (OR) = 0.67, 95% CI 2-sided [0.30 to 1.53], Standard Error of Mean .28 — Odds of believing VLNC are less harmful than cigarettes in the Nicotine corrective with reason for misperception/odds of believing VLNC are less harmful than cigarettes in the condition with both component of coherence
Statistical Analysis 4: Comparison: Nicotine Corrective Control vs Nicotine Corrective With Both Components of Coherence; Adjusted logistic regression showing the effect of condition (Nicotine corrective control compared to the Nicotine corrective with both components of coherence (reference group)) on VLNC relative harm beliefs controlling for baseline beliefs and VLNC use; Test type: Superiority; p = 0.360, Regression, Logistic; Odds Ratio (OR) = 1.56, 95% CI 2-sided [0.60 to 4.04], Standard Error of Mean .76 — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 5: Comparison: Nicotine Corrective With Causal Explanation vs Nicotine Corrective With Both Components of Coherence; Adjusted logistic regression showing the effect of condition (Nicotine corrective with causal explanation compared to the Nicotine corrective with both components of coherence (reference group)) on VLNC relative harm beliefs controlling for baseline beliefs and VLNC use; Test type: Superiority; p = 0.765, Regression, Logistic; Odds Ratio (OR) = 1.14, 95% CI 2-sided [0.48 to 2.70], Standard Error of Mean .50 — [estimate comment as in outcome 4, analysis 2]
Statistical Analysis 6: Comparison: Nicotine Corrective With Reason for Misperception vs Nicotine Corrective With Both Components of Coherence; Adjusted logistic regression showing the effect of condition (Nicotine corrective with reason for misperception compared to the Nicotine corrective with both components of coherence (reference group)) on VLNC relative harm beliefs controlling for baseline beliefs and VLNC use; Test type: Superiority; p = 0.252, Regression, Logistic; Odds Ratio (OR) = 0.60, 95% CI 2-sided [0.25 to 1.43], Standard Error of Mean .27 — [estimate comment as in outcome 4, analysis 3]

5. Primary Outcome: Change in Inferential Beliefs Regarding Smokeless Tobacco
Description: Participants will be shown a written description of smokeless tobacco before answering questions about them: "The next questions are about smokeless tobacco. Smokeless tobacco like chewing, oral, or spit tobacco come as loose leaves, plugs, or twists of dried tobacco that may be flavored. It's chewed or placed between the cheek and gum or teeth. The user spits out (or swallows) the saliva that has soaked through the tobacco. Dissolvables are another type of product that dissolves in the mouth and can be sold as lozenges, strips, or sticks. Nicotine is absorbed through the mouth tissues." Participants will also see a picture of these products with the description. Response options were dichotomized to low relative harm perceptions (much less harmful, somewhat less harmful) and high relative harm perceptions (much more harmful, somewhat more harmful, not less or more harmful).
Time Frame: Baseline and up to 5 minutes after receiving the corrective message
Measure: Count of Participants; unit: Participants
Arm/Group | Nicotine Corrective Control | Nicotine Corrective With Causal Explanation | Nicotine Corrective With Reason for Misperception | Nicotine Corrective With Both Components of Coherence
Number analyzed (Participants) | 42 | 53 | 56 | 42
Participants
  Low relative harm perception | 17 | 32 | 22 | 26
  High relative harm perception | 22 | 20 | 31 | 15
  Missing | 3 | 1 | 3 | 1
Statistical Analysis 1: Comparison: Nicotine Corrective Control vs Nicotine Corrective With Both Components of Coherence; Unadjusted logistic regression showing the effect of condition (Nicotine corrective control compared to the Nicotine corrective with both components of coherence (reference group)) on smokeless tobacco relative harm beliefs; Test type: Superiority; p = 0.077, Regression, Logistic; Odds Ratio (OR) = 0.45, 95% CI 2-sided [0.18 to 1.09], Standard Error of Mean .20 — Odds of believing smokeless tobacco is less harmful than cigarettes in the control condition/odds of believing smokeless tobacco is less harmful than cigarettes in the condition with both component of coherence
Statistical Analysis 2: Comparison: Nicotine Corrective With Causal Explanation vs Nicotine Corrective With Both Components of Coherence; Unadjusted logistic regression showing the effect of condition (Nicotine corrective with causal explanation compared to the Nicotine corrective with both components of coherence (reference group)) on smokeless tobacco relative harm beliefs; Test type: Superiority; p = 0.853, Regression, Logistic; Odds Ratio (OR) = 0.92, 95% CI 2-sided [0.40 to 2.15], Standard Error of Mean .40; Odds of believing smokeless tobacco is less harmful than cigarettes in the Nicotine corrective with causal explanation/odds of believing smokeless tobacco is less harmful than cigarettes in the condition with both component of coherence
Statistical Analysis 3: Comparison: Nicotine Corrective With Reason for Misperception vs Nicotine Corrective With Both Components of Coherence; Unadjusted logistic regression showing the effect of condition (Nicotine corrective with reason for misperception compared to the Nicotine corrective with both components of coherence (reference group)) on smokeless tobacco relative harm beliefs; Test type: Superiority; p = 0.037, Regression, Logistic; Odds Ratio, log = 0.41, 95% CI 2-sided [0.18 to 0.95], Standard Error of Mean .18 — Odds of believing smokeless tobacco is less harmful than cigarettes in the Nicotine corrective with both components of coherence/odds of believing smokeless tobacco is less harmful than cigarettes in the condition with both component of coherence
Statistical Analysis 4: Comparison: Nicotine Corrective Control vs Nicotine Corrective With Both Components of Coherence; Adjusted logistic regression showing the effect of condition (Nicotine corrective control compared to the Nicotine corrective with both components of coherence (reference group)) on smokeless relative harm beliefs controlling for baseline beliefs and smokeless tobacco use; Test type: Superiority; p = 0.349, Regression, Logistic; Odds Ratio (OR) = 0.60, 95% CI 2-sided [0.21 to 1.75], Standard Error of Mean .33 — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 5: Comparison: Nicotine Corrective With Causal Explanation vs Nicotine Corrective With Both Components of Coherence; Adjusted logistic regression showing the effect of condition (Nicotine corrective with causal explanation compared to the Nicotine corrective with both components of coherence (reference group)) on smokeless relative harm beliefs controlling for baseline beliefs and smokeless tobacco use; Test type: Superiority; p = 0.464, Regression, Logistic; Odds Ratio (OR) = 1.45, 95% CI 2-sided [0.54 to 3.93], Standard Error of Mean .74 — Odds of believing smokeless tobacco is less harmful than cigarettes in the Nicotine corrective with causal explanation/odds of believing smokeless tobacco is less harmful than cigarettes in the condition with both component of coherence
Statistical Analysis 6: Comparison: Nicotine Corrective With Reason for Misperception vs Nicotine Corrective With Both Components of Coherence; Adjusted logistic regression showing the effect of condition (Nicotine corrective with reason for misperception compared to the Nicotine corrective with both components of coherence (reference group)) on smokeless relative harm beliefs controlling for baseline beliefs and smokeless tobacco use; Test type: Superiority; p = 0.187, Regression, Logistic; Odds Ratio (OR) = 0.50, 95% CI 2-sided [0.18 to 1.40], Standard Error of Mean .26 — Odds of believing smokeless tobacco is less harmful than cigarettes in the Nicotine corrective with reason for misperception/odds of believing smokeless tobacco is less harmful than cigarettes in the condition with both component of coherence

6. Primary Outcome: Change in Inferential Beliefs Regarding Cigarillos
Description: Participants will be shown a written description of smokeless tobacco before answering questions about them: "The next questions are about cigarillos. Cigarillos look like small versions of traditional cigars, but can be bought in packages of one or two. Cigarillos smoke is often inhaled, unlike cigar smoke which is often held in the mouth and then released. Cigarillos are often flavored. Swisher Sweets, White Owl, and Dutch Masters are common cigarillo brands.." Participants will also see a picture of these products with the description. Response options were dichotomized to low relative harm perceptions (much less harmful, somewhat less harmful) and high relative harm perceptions (much more harmful, somewhat more harmful, not less or more harmful).
Time Frame: Baseline and up to 5 minutes after receiving the corrective message
Measure: Count of Participants; unit: Participants
Arm/Group | Nicotine Corrective Control | Nicotine Corrective With Causal Explanation | Nicotine Corrective With Reason for Misperception | Nicotine Corrective With Both Components of Coherence
Number analyzed (Participants) | 42 | 53 | 56 | 42
Participants
  Low relative harm perception | 6 | 5 | 6 | 6
  High relative harm perception | 33 | 44 | 49 | 35
  Missing | 3 | 4 | 1 | 1
Statistical Analysis 1: Comparison: Nicotine Corrective Control vs Nicotine Corrective With Both Components of Coherence; Unadjusted logistic regression showing the effect of condition (Nicotine corrective control compared to the Nicotine corrective with both components of coherence (reference group)) on cigarillo relative harm beliefs; Test type: Superiority; p = 0.925, Regression, Logistic; Odds Ratio (OR) = 1.06, 95% CI 2-sided [0.31 to 3.62], Standard Error of Mean .66 — Odds of believing cigarillos are less harmful than cigarettes in the control condition/odds of believing cigarillos are less harmful than cigarettes in the condition with both component of coherence
Statistical Analysis 2: Comparison: Nicotine Corrective With Causal Explanation vs Nicotine Corrective With Both Components of Coherence; Unadjusted logistic regression showing the effect of condition (Nicotine corrective with causal explanation compared to the Nicotine corrective with both components of coherence (reference group)) on cigarillo relative harm beliefs; Test type: Superiority; p = 0.525, Regression, Logistic; Odds Ratio (OR) = 0.66, 95% CI 2-sided [0.19 to 2.35], Standard Error of Mean .43 — Odds of believing cigarillos are less harmful than cigarettes in the Nicotine corrective with causal explanation/odds of believing cigarillos are less harmful than cigarettes in the condition with both component of coherence
Statistical Analysis 3: Comparison: Nicotine Corrective With Reason for Misperception vs Nicotine Corrective With Both Components of Coherence; Unadjusted logistic regression showing the effect of condition (Nicotine corrective with reason for misperception compared to the Nicotine corrective with both components of coherence (reference group)) on cigarillo relative harm beliefs; Test type: Superiority; p = 0.586, Regression, Logistic; Odds Ratio (OR) = 0.71, 95% CI 2-sided [0.21 to 2.40], Standard Error of Mean .44 — Odds of believing cigarillos are less harmful than cigarettes in the Nicotine corrective with reason for misperception/odds of believing cigarillos are less harmful than cigarettes in the condition with both component of coherence
Statistical Analysis 4: Comparison: Nicotine Corrective Control vs Nicotine Corrective With Both Components of Coherence; Adjusted logistic regression showing the effect of condition (Nicotine corrective control compared to the Nicotine corrective with both components of coherence (reference group)) on cigarillo relative harm beliefs controlling for smokeless tobacco use; Test type: Superiority; p = 0.883, Regression, Logistic; Odds Ratio (OR) = 1.10, 95% CI 2-sided [0.31 to 3.90], Standard Error of Mean .71 — [estimate comment as in outcome 6, analysis 1]
Statistical Analysis 5: Comparison: Nicotine Corrective With Causal Explanation vs Nicotine Corrective With Both Components of Coherence; Adjusted logistic regression showing the effect of condition (Nicotine corrective with causal explanation compared to the Nicotine corrective with both components of coherence (reference group)) on cigarillo relative harm beliefs controlling for smokeless tobacco use; Test type: Superiority; p = 0.534, Regression, Logistic; Odds Ratio (OR) = 0.66, 95% CI 2-sided [0.18 to 2.41], Standard Error of Mean .44 — [estimate comment as in outcome 6, analysis 2]
Statistical Analysis 6: Comparison: Nicotine Corrective With Reason for Misperception vs Nicotine Corrective With Both Components of Coherence; Adjusted logistic regression showing the effect of condition (Nicotine corrective with reason for misperception compared to the Nicotine corrective with both components of coherence (reference group)) on cigarillo relative harm beliefs controlling for smokeless tobacco use; Test type: Superiority; p = 0.661, Regression, Logistic; Odds Ratio (OR) = 0.76, 95% CI 2-sided [0.22 to 2.62], Standard Error of Mean .48 — [estimate comment as in outcome 6, analysis 3]

7. Primary Outcome: Change in Beliefs About Intention to Switch Products
Description: The extent to which participants agree or disagree with the following statement: I would consider completely switching to a tobacco product that is not lit on fire rather than continuing to smoke cigarettes. Response options are a continuous scale from 0 "I do not agree at all" to 100, "I completely agree."
Time Frame: Baseline and up to 5 minutes after receiving the corrective message
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Nicotine Corrective Control | Nicotine Corrective With Causal Explanation | Nicotine Corrective With Reason for Misperception | Nicotine Corrective With Both Components of Coherence
Number analyzed (Participants) | 42 | 53 | 56 | 42
units on a scale | 60.6 (30.3) | 53.5 (36.4) | 56.4 (34.3) | 57.9 (34.4)
Statistical Analysis 1: Comparison: Nicotine Corrective Control vs Nicotine Corrective With Both Components of Coherence; ANCOVA adjusted for baseline consideration of switching; Test type: Superiority; p = 0.965, ANCOVA; Sidak's adjusted p-value (df=4); Mean Difference (Final Values) = 1.97, 95% CI 2-sided [-9.25 to 13.19], Standard Error of Mean 4.66 — Nicotine corrective control - Nicotine corrective with both components of coherence
Statistical Analysis 2: Comparison: Nicotine Corrective With Causal Explanation vs Nicotine Corrective With Both Components of Coherence; ANCOVA adjusted for baseline consideration of switching; Test type: Superiority; p = 0.979, ANCOVA; Sidak's adjusted p-value (df=4); Mean Difference (Final Values) = 1.57, 95% CI 2-sided [-9.13 to 12.27], Standard Error of Mean 4.44; Nicotine corrective with causal explanation - Nicotine corrective with both components of coherence
Statistical Analysis 3: Comparison: Nicotine Corrective With Reason for Misperception vs Nicotine Corrective With Both Components of Coherence; ANCOVA adjusted for baseline consideration of switching; Test type: Superiority; p = 0.73, ANCOVA; Sidak's adjusted p-value (df=4); Mean Difference (Final Values) = 4.07, 95% CI 2-sided [-6.46 to 14.59], Standard Error of Mean 4.37; Nicotine corrective with reason for misperception - Nicotine corrective with both components of coherence

ADVERSE EVENTS:
Time Frame: up to 3 months
Arm/Group | Nicotine Corrective Control | Nicotine Corrective With Causal Explanation | Nicotine Corrective With Reason for Misperception | Nicotine Corrective With Both Components of Coherence
All-Cause Mortality (participants affected / at risk) | 0/42 | 0/53 | 0/56 | 0/42
Serious Adverse Events (participants affected / at risk) | 0/42 | 0/53 | 0/56 | 0/42
Other Adverse Events (participants affected / at risk) | 0/42 | 0/53 | 0/56 | 0/42

LIMITATIONS AND CAVEATS:
Smokers on MTurk are unlikely to be representative of US smokers. The nicotine misperception was measured on a continuous 0-100 scale and was able to detect smaller changes than the dichotomous relative harm perception outcome. Participants who reported believing nicotine causes cancer may accurately understand that nicotine indirectly causes disease because it keeps people exposed to carcinogens over time, resulting in misclassification.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-08-04): https://cdn.clinicaltrials.gov/large-docs/92/NCT05129592/Prot_SAP_000.pdf